CLINICAL TRIAL: NCT05232162
Title: Establishment of Reference Ranges for Aldosterone and Renin in a Multi-racial Community Using the Chemiluminescent Immunoassay (CLIA)
Brief Title: Establishment of Aldosterone and Renin Reference Range
Acronym: ARR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Malaysia Sarawak (Other)
Responsible Party: Sponsor
Other Study IDs: ARR reference range
Record Dates: First submitted 2022-01-30; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Aldosteronism
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Elevated aldosterone levels were also shown to contribute to the excess morbidity and mortality. Literature shows aldosterone and renin levels differ between ethnicity and gender. There is no established reference intervals for these two hormone levels in Asian community. We aim to establish reference intervals for plasma aldosterone and direct renin concentrations among Malaysians residing in Sarawak using the chemiluminescent immunoassay (CLIA).

This is a cross-sectional study which will be conducted among ambulatory patients, healthy blood donors and healthy volunteers. 300 participants who fulfil study criteria will be recruited after informed consent.

Socio-demographic data and anthropometric measurements will be recorded. Blood will be taken for plasma aldosterone, renin, serum potassium and creatinine. Urine will be collected for estimation of 24-hour sodium excretion. Aldosterone and renin reference intervals will be established partitioned for gender.

DETAILED DESCRIPTION:
Despite old beliefs that Primary Aldosteronism (PA) is uncommon and warrants screening only when patients present with hypertension and hypokalemia, it is now believed that PA is in fact the most common cause of secondary hypertension, accounting for 5-13% of the hypertensive cohort, with an even higher prevalence among those with resistant hypertension. This stems from more efficient screening of this condition with the widespread use of the aldosterone to renin ratio. It is a disorder in which the adrenal cortex autonomously produces excessive aldosterone leading to sodium and water retention, resulting in a subsequent rise of blood pressure (BP), and down-regulation of renin through the renin-angiotensin-aldosterone system (RAAS) pathway.

Once considered a relatively benign condition, PA has been unequivocally shown to have effects beyond its effects on BP levels. Hypertension alone could not explain the higher adverse cardiovascular outcomes as PA patients were found to have higher cardiovascular mortality compared to patients with essential hypertension (EH) despite being matched for cardiovascular risks.

Elevated aldosterone levels were also shown to contribute to the excess morbidity and mortality. Recent studies have shown that PA is associated with a myriad of other co-morbidities, particularly cardiovascular and renal injuries, which might play a role in contributing to the elevated morbidity and mortality.

Traditionally, the activity of renin-angiotensin-aldosterone system is evaluated by measurement of plasma renin activity (PRA). However, PRA measurement is a complex procedure with poor inter-laboratory reproducibility, which makes it a limitation preventing more extensive use of PRA for diagnostic purposes. Direct renin assay is a new chemiluminescent renin assay, which utilizes the high specificity of monoclonal antibodies to detect the renin molecule, and is proven as a good alternative to the use of PRA. The use of this new assay appears to be simpler, faster and more reproducible than PRA, which is shown in a recent multi-center comparative study.

Literature shows aldosterone and renin levels differ between ethnicity and gender. There is no established reference intervals for these two hormone levels in Asian community.

General objective:

To establish reference intervals for plasma aldosterone and direct renin concentrations among Asians in the Sarawak population using the chemiluminescent immunoassay (CLIA).

Specific objective:

To compare reference ranges among gender.

This is a cross-sectional study which will be conducted among ambulatory patients, healthy blood donors and healthy volunteers. Participants who fulfil study criteria will be recruited after informed consent.

The inclusion criteria are subjects who are:

1. aged 18 years old and above
2. agreeable to participate in this study
3. Malaysian
4. normal kidney function (eGFR>60ml/min/1.73m2)
5. BMI<27.5kg/m2

Whereas exclusion criteria are subjects who are

1. taking prescribed/OTC medications within 3 months of study
2. taking estrogen, either oral contraceptive pills or hormone replacement therapy
3. having hypertension defined as systolic blood pressure>140 and/or diastolic blood pressure>90mmHg or on anti-hypertensive
4. pregnant
5. smokers

Socio-demographic data on age, gender, ethnicity, body mass index (BMI), medication usage, smoking and pregnancy status will be recorded. Seated blood pressure will be measured using appropriately-sized cuff after 5 minutes of rest. The mean of 2 readings will be recorded.

A total of 10ml of whole blood will be withdrawn after the subjects have been seated for at least 15 minutes, between 8am and 10am. Blood drawn will be collected into appropriate specimen tubes - potassium EDTA tubes for plasma aldosterone and plasma renin; plain tubes for measurement of serum potassium and creatinine. Urine will be collected for estimation of 24-hour sodium excretion.

Specimen tubes will be kept at room temperature and transported within 30 minutes of blood drawn to the laboratory for immediate processing (centrifugation, separation and freezing of plasma). Plasma will be stored in a temperature-controlled freezer at -20C for a maximum of six months prior to analysis on the Liaison instrument. Measurements of plasma aldosterone will be performed using chemiluminescent immunoassay (CLIA) aldosterone kit (DiaSorin S.p.A., Italy), with inter-assay and intra-assay coefficient variations (CV) of less than 10% and 4.2% respectively. Measurements of plasma renin will be done using chemiluminescent immunoassay (CLIA) renin kit (DiaSorin S.p.A., Italy). Serum potassium and creatinine will be processed within 2 hours of blood draw. The samples will be stored for a maximum of two weeks prior to analysis. The eGFR will be calculated using the Modification of Diet in Renal Disease (MDRD) Study equation. Urine will be stored for a maximum of two weeks prior to analysis for urine sodium, potassium and creatinine. Sodium excretion will be calculated using INTERSALT formula.

The participation duration for each participant is 30 minutes.

Withdrawal criteria Participants can choose to withdraw at any time after informed consent. Participants may be withdrawn if the investigator deems that it is unsuitable for the participants to be involved in this study. Withdrawn participants will be replaced until sample size is adequate.

Sample size We aim to recruit 300 participants (150 males and 150 females) for the purpose of establishing the reference interval of aldosterone and renin among Malaysians residing in Sarawak.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years old and above
2. agreeable to participate in this study
3. normal kidney function (eGFR>60ml/min/1.73m2)
4. Malaysian
5. BMI<27.5kg/m2

Exclusion Criteria:

1. taking prescribed/OTC medications within 3 months of study
2. taking estrogen, either in oral contraceptive pills or hormone replacement therapy
3. having hypertension defined as blood pressure>140/90mmHg or on anti-hypertensive
4. having hypokalemia (serum potassium <3.5mmol/L)
5. pregnant
6. smoker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Ambulatory healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Aldosterone and renin reference intervals | 24 months

SECONDARY OUTCOMES:
Aldosterone and renin reference intervals partitioned for gender | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Malaysia Sarawak, Kuching, Sarawak, Malaysia

IPD SHARING:
Plan to Share IPD: No